CLINICAL TRIAL: NCT02455492
Title: An Epidemiological Investigation Into the Association Between Recent Stroke, Acute Coronary Syndrome or Pneumonia and Adverse Perioperative Outcomes Following Elective Non-cardiac and Cardiac Surgery
Brief Title: Factors Associated With Perioperative Outcomes in Non-emergency Surgery
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 15_034R
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Stroke; Acute Coronary Syndrome; Pneumonia
Keywords: Mortality; Perioperative period; Elective surgical procedures
MeSH Terms: conditions — Stroke; Acute Coronary Syndrome; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: stroke or myocardial infarction or pneumonia — There are three main exposure groups with exposure defined as a binary variable (yes/no): Stroke in the six months prior to surgery; Myocardial infarction in the six months prior to surgery; Pneumonia in the six months prior to surgery

SUMMARY:
This epidemiological study investigates the association of recent stroke, acute coronary syndrome or pneumonia and adverse perioperative outcomes following elective non-cardiac and cardiac surgery using routinely collected UK primary and secondary care patient data.

DETAILED DESCRIPTION:
Previous studies have identified prior stroke, heart attack or current diabetes mellitus and anaemia as important risk factors for adverse outcomes following surgery. Recent heart attacks are associated with greater risks than older ones. While recent data suggests that newer strokes impart significantly greater risk than older strokes, there is a lack of concordance on the literature on this, despite the plausibility of the finding. Despite knowledge that prior pneumonia has long-term health risks, there is a lack of data on whether prior pneumonia influences perioperative risk or whether the time interval from pneumonia to surgery affects this relationship. Furthermore while diabetes mellitus and anaemia are known to be important perioperative risk factors, the relationship between haemoglobin concentration or HbA1c levels and perioperative outcomes is unclear. The aim of this epidemiological study is to explore these associations with perioperative risk in the United Kingdom Clinical Practice Research Datalink (with linkage to Hospital Episode Statistics data and Office of National Statistics mortality data).

The research aims are:

1. To investigate the association between three recent acute medical events (stroke, pneumonia and MI) and adverse perioperative outcomes following non-cardiac and cardiac surgery.
2. To investigate the association between time-elapsed between acute medical events (stroke, pneumonia and MI) and adverse perioperative outcomes following non-cardiac and cardiac surgery.
3. To investigate numerical risk thresholds for haemoglobin and HbA1c that could predict adverse perioperative outcomes following non-cardiac and cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergone a non-cardiac or cardiac elective procedure between 1/01/2004 and 31/12/2013

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients within the Clinical Practice Research Datalink who have undergone a non-cardiac or cardiac elective procedure between 1/01/2004 and 31/12/2013.
Sampling Method: Probability Sample
Enrollment: 266436 (Actual)
Dates: Start 2004-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Perioperative mortality (yes/no) | up to 60 days of surgery
  all-cause mortality within the specified time frame; both in and out of hospital; as recorded in primary care patient record and validated using Office of National Statistics death certification records; unadjusted and adjusted relative risks will be calculated (odds ratios and hazard ratios)

SECONDARY OUTCOMES:
Acute coronary syndrome (yes/no) | within 30 days of surgery
  physician diagnosed and occurring within the specified time frame; as recorded in patient care record; unadjusted and adjusted relative risks will be calculated (odds ratios and hazard ratios)
Pneumonia (yes/no) | within 30 days of surgery
  physician diagnosed and occurring within the specified time frame; as recorded in patient care records; unadjusted and adjusted relative risks will be calculated (odds ratios and hazard ratios)

CONTACTS AND LOCATIONS:
Overall Officials: Puja R Myles, PhD, Study Director — University of Nottingham